CLINICAL TRIAL: NCT05787522
Title: Prospective, Multicenter, Randomized Evaluation of the Performance and Clinical Applicability of AI-Assisted Radiotherapy Contouring Software for Thoracic Organs at Risk
Brief Title: Clinical Validation of AI-Assisted Radiotherapy Contouring Software for Thoracic Organs at Risk
Status: Completed | Type: Observational
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Collaborators: Guangzhou Perception Vision Medical Technology Co. Ltd (Unknown); People's Hospital of Guangxi Zhuang Autonomous Region (Other); Shanxi Province Cancer Hospital (Other); Fifth Affiliated Hospital, Sun Yat-Sen University (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor
Other Study IDs: PVMEDCT202201
Record Dates: First submitted 2023-03-02; First posted 2023-03-28 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Lung Cancer; Breast Cancer; Esophageal Cancer
Keywords: Artificial Intelligence; Radiotherapy; contouring; thoracic organs at risk
MeSH Terms: conditions — Lung Neoplasms; Breast Neoplasms; Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Independent manual contouring: Manual contouring refers to physicians using the brush tool on the contouring platform to segment thoracic organs at risk manually, without the use of auto-segmentation tools.
- AI contouring: AI contouring refers to the auto-segmentation results generated by the Res-SE Net model, with the model integrated into the auto-segmentation software (iCurveE).
- AI-assisted contouring: After generating the AI contouring results, investigators will import them into the contouring platform and perform manual modifications, producing the AI-assisted contouring.

SUMMARY:
The goal of this clinical trial is to evaluate performance and clinical applicability of AI-assisted radiotherapy contouring software (iCurveE) for thoracic organs at risk. The main question it aims to answer is:

• Does AI-assisted contouring (AI contouring with manual modification) offer greater accuracy and time efficiency compared to manual contouring? After screening, the qualified participants' thoracic CT images will be anonymized and segmented using three methods: manual, AI (AI-only), and AI-assisted contouring. The researchers will compare the results generated by the three different contouring methods with the ground truth established by expert consensus, in order to evaluate both accuracy and time-related parameters

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years old, no gender limit.
2. Patients diagnosed with breast cancer, lung cancer, or esophageal cancer, who are scheduled for chest CT scanning followed by thoracic radiotherapy.
3. CT slice thickness ≤5mm.
4. Patients understand the goal of the trial, are willing to attend the trial and sign the informed consent.

Exclusion Criteria:

1. Congenital malformations or abnormal anatomical structures resulting from non-tumor factors in the scan area.
2. Artifact, prosthesis or implantation causing images undistinguishable.
3. CT images not conforming to DICOM standards.
4. Investigators consider not suitable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This trial will enroll 500 patients with lung, esophageal, or breast cancer, who are scheduled to receive thoracic radiotherapy across five clinical cancer institutes.
Sampling Method: Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2022-09-30 (Actual); Primary Completion 2023-07-27 (Actual); Study Completion 2024-03-06 (Actual)

PRIMARY OUTCOMES:
volumetric DICE similarity coefficient, vDSC | Within 6 months after enrollment
  vDSC= 2×（A∩B）/(A+B), where A refers to the volume of the ground truth, and B refers to the volume of the manual, AI, or AI-assisted contour.
Contouring time (min) | Within 6 months after enrollment
  Manual contouring time is recorded from the time the CT is loaded on the contouring platform to the completion of contouring. AI-assisted contouring time is defined as the sum of the auto-segmentation model runtime, the transfer to the contouring platform, and the subsequent manual modification.

SECONDARY OUTCOMES:
95th percentile Hausdorff Distance, HD95 | Within 6 months after enrollment
  HD95(A, B) = max (h95(A, B), h95(B, A)), where h95(A, B) is the 95th percentile of the shortest distances from all points on surface A to surface B, and vice-versa for h95(B, A). A represents the ground truth and B represents the manual, AI or AI-assisted delineation
Surface DICE similarity coefficient, sDSC | Within 6 months after enrollment
  sDSC = (|S(A) ∩ S(B)τ| + |S(B) ∩ S(A)τ|) / (|S(A)| + |S(B)|), where S(A) and S(B) are the sets of points on the surfaces of A and B, S(B)τ represents the points on surface B that are within the tolerance τ of surface A, and S(A)τ represents the points on surface A that are within the tolerance τ of surface B. A represents the ground truth and B represents the manual, AI or AI-assisted delineation
Rate of time efficiency improvement | Within 6 months after enrollment
  Rate of efficiency time improvement= (manual contouring duration - AI-assisted contouring duration)/ manual contouring duration*100%
Volumetric revision index, VRI | Within 6 months after enrollment
  VRI = [(A- A∩B) + (B- A∩B)] /A, where A refers to the volume of the ground truth, and B refers to the volume of the manual, AI, or AI-assisted contour.
Recall, Rec | Within 6 months after enrollment
  Rec = | A∩B| / A, where A refers to the volume of the ground truth, and B refers to the volume of the manual, AI, or AI-assisted contour.
Precision, Pre | Within 6 months after enrollment
  Pre= |A∩B| / B, where A refers to the volume of the ground truth, and B refers to the volume of manual, AI, or AI-assisted contour.
Relative volume difference, RVD | Within 6 months after enrollment
  RVD = |A-B| /A, where A refers to the volume of the ground truth, and B refers to the volume of the manual, AI, or AI-assisted contour.
Investigators satisfaction score for AI contouring | Within 6 months after enrollment
  Evaluated on a 1-5 Likert scale: 1 - strongly dissatisfied, 2 - dissatisfied, 3 - neutral, 4 - satisfied, 5 - strongly satisfied.

OTHER OUTCOMES:
Number of adverse events, AEs | Within 1 day after CT scanning
  Participant Adverse events during CT scanning
Number of device defects during AI-assisted contouring | Within 6 months after enrollment
  Number of failures in generating, transferring, or saving auto-segmentation results

CONTACTS AND LOCATIONS:
Overall Officials: Zhiyong Yuan, Ph.D., Principal Investigator — Tianjin Medical University Cancer Institute and Hospital
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin Key Laboratory of Cancer Prevention and Therapy, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
The protocol of this study are available from the corresponding author upon reasonable request after the manuscript publication.
Supporting Information: Study Protocol
Time Frame: Beginning 1 year after publication with no end date.
Access Criteria: Requests must include a detailed protocol, analysis plan, and data exchange with institutional approvals in place before data transfer of any information.